CLINICAL TRIAL: NCT07110038
Title: DEPECA-1 - DEfeating PEnile Cancer 1 - A Phase II Study to Evaluate a First-line Systemic Therapy With Enfortumab Vedotin Plus Avelumab for Advanced and Metastatic Penile Carcinoma
Brief Title: DEPECA-1 - A Phase II Study to Evaluate a First-line Systemic Therapy With Enfortumab Vedotin Plus Avelumab for Advanced and Metastatic Penile Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry); Astellas Pharma GmbH (Industry); University Hospital Tübingen (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UKT-IKF-DEPECA-1; 2025-521644-37-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-18; First posted 2025-08-07 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Penile Squamous Cell Carcinoma (PSCC)
MeSH Terms: interventions — avelumab; enfortumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined therapy consisting of enfortumab vedotin and avelumab (Experimental)
  Interventions: Drug: Avelumab; Drug: enfortumab vedotin

INTERVENTIONS:
Drug: Avelumab — Avelumab, 1,200 mg IV
Drug: enfortumab vedotin — Enfortumab vedotin, 1.25 mg/kg IV

SUMMARY:
The DEPECA-1 trial is the first systematic Phase II trial to evaluate response and survival to a combination of antibody-drug conjugate enfortumab vedotin plus the PD-L1 inhibitor avelumab in patients with locally advanced and metastatic penile squamous cell carcinoma (PeCa) in the 1st line setting.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has ability to understand and the willingness to sign a written informed consent.
2. Patient is ≥ 18 years of age at time of signing the written informed consent.
3. Male patients with histologically confirmed diagnosis of penile squamous cell carcinoma.
4. Patients must be considered non-eligible for curative surgical management. Eligibility for trial inclusion should be based on the presence of either distant metastatic disease (M1) or at least one of the following scenarios based on the UICC/AJCC 8th edition TNM clinical and pathological classification of penile cancer:

   1. Stage 3 (cT3) disease with a single lymph node involved (N1).
   2. Stage 4 disease (cT4).
   3. Any T stage with either N2 (involvement of multiple or bilateral inguinal nodes) or N3 (fixed inguinal nodal mass or pelvic lymphadenopathy) disease. Patients without distant metastases are eligible if multidisciplinary team review concludes that they are unsuitable for curative surgery.
5. Tumor material (archival or current) is available for local pathology testing (PD-L1, HPV).
6. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
7. Measurable disease per RECIST 1.1 criteria.
8. No prior systemic therapy for metastatic or locally advanced PeCa in the palliative setting. NOTE: (Neo)adjuvant systemic therapy (without IO) is allowed at least 6 months before study enrollment.
9. Patients has adequate blood count, liver-enzymes, and renal function:

   1. ANC (Absolute neutrophil count) > 1,500 cells/μL without the use of hematopoietic growth factors.
   2. Platelet count ≥ 100 x 109/L (>100,000 per mm3).
   3. Hemoglobin ≥ 9 g/dL.
   4. Serum total bilirubin ≤ 1.5x institutional upper normal limit (ULN).
   5. AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional ULN (or ≤ 5 x ULN if liver metastases are present).
   6. Creatinine clearance ≥ 30 mL/min as calculated by the Cockcroft- Gault equation (or local institutional standard method).
10. No other active malignancy within the past 3 years, except for adequately treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin.
11. No history of significant cardiovascular disease (e.g., myocardial infarction, unstable angina) within the last 6 months.
12. Life expectancy of at least 3 months.
13. Willingness to comply with study requirements, including follow-up visits and procedures.
14. Patients with female partners of childbearing potential must agree to use an effective method of contraception during the study and for 4 months after the last dose of enfortumab vedotin or for at least 30 days after last avelumab treatment administration, whichever occurs last.

Exclusion Criteria:

1. Previous systemic therapy for metastatic or locally advanced PeCa in the palliative setting.
2. Previous treatment with investigational drugs or devices within 30 days prior to the first dose of trial treatment.
3. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
4. Active, known, or suspected autoimmune disease requiring systemic treatment within the past 2 years. Patients with controlled autoimmune d disease not requiring systemic immunosuppressive treatment including diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases are eligible.
5. Has ongoing sensory or motor neuropathy Grade 2 or higher.
6. Has a history of uncontrolled diabetes (HbA1c > 8%).
7. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
8. Active infection requiring systemic therapy. The following exceptions apply:

   1. Patients with an HIV infection are eligible if they are on effective antiretroviral therapy with undetectable viral load within 6 months, provided there is no expected drug-drug interaction.
   2. Patients with evidence of chronic HBV infection are eligible if the HBV viral load is undetectable on suppressive therapy (if indicated), and if they have ALT, AST, and total bilirubin levels < ULN, and provided there is no expected drug-drug interaction.
   3. Patients with a history of HCV infection are eligible if they have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load, and if they have ALT, AST, and total bilirubin levels < ULN.
9. History of other malignancies within the past 3 years, with the exception of adequately treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin.
10. Severe hepatic impairment (Child-Pugh Class C).
11. Severe renal impairment or requirement for dialysis.
12. History of keratitis and corneal ulceration in the last two years.
13. Active pneumonia, pneumonitis or pulmonary fibrosis.
14. Active tuberculosis.
15. Known prior severe hypersensitivity to the study drugs or any component of their formulations, known severe hypersensitivity reactions to monoclonal antibodies (NCT CTCAE Grade ≥ 3).
16. Inability or unwillingness to comply with study requirements, including follow-up visits and procedures.
17. Inability to provide informed consent.
18. Use of immunosuppressive medication within 14 days prior to the first dose of study treatment, with the exception of intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra-articular injection), systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent, or steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
19. Prior organ transplantation including allogenic stem-cell transplantation.
20. Vaccination within 4 weeks of the first dose of avelumab and while on trials is prohibited except for administration of inactivated vaccines.
21. Persisting toxicity related to prior therapy (NCI CTCAE Grade > 1); however, alopecia or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.
22. Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
23. Patient participated in another interventional clinical study according to Medicines Act within 28 days prior to study enrollment or participation in a clinical study according to Medicines Act at the same time as this study unless it is an observational / non-interventional study or during the follow- up period of an interventional study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 24 months.
  Objective Response Rate (ORR) in 1st line as assessed by investigators, defined as the proportion of patients achieving a complete response (CR) or partial response (PR) according to RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 5 years.
  Progression-free survival (PFS), defined as the time from the start of treatment to the first documented disease progression acc. to RECIST 1.1 criteria or death from any cause, whichever occurs first.
Overall Survival (OS) | Up to 5 years.
  Time from the start of treatment to death from any cause.
Duration of Response (DoR) | Up to 5 years.
  Time from the first documented response (CR or PR) to disease progression or death from any cause (whichever occurs first).
Disease Control Rate (DCR) | Up to 27 months.
  Disease Control Rate (DCR), defined as the proportion of patients achieving CR, PR, or stable disease (SD) for at least 12 weeks according to RECIST 1.1 criteria.
Incidence and severity of (serious) adverse events | Up to 27 months
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Quality of life (QoL) using EQ-5D-5L questionnaire | Up to 24 months.
  Changes in patient-reported quality of life, using EQ-5D-5L questionnaire and a set of bolt-on questions will be collected.
Quality of life (QoL) using EQ-HWB-S questionnaire | Up to 24 months.
  Changes in patient-reported quality of life, using EQ-HWB-S questionnaire and a set of bolt-on questions will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof. Dr., Study Chair — Frankfurter Institut für Klinische Krebsforschung IKF GmbH
Locations (2):
- Germany (2):
  - University Hospital Mannheim, Mannheim
  - University Hospital Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: No